CLINICAL TRIAL: NCT06126692
Title: 3TR Asthma Biologics Cohort (ABC) Study - A Part of the 3TR (Taxonomy, Treatment, Targets and Remission) Consortium for the Identification of the Molecular Mechanisms of Non-response to Treatment, Relapses, and Remission in Autoimmune, Inflammatory, and Allergic Conditions
Brief Title: 3TR Asthma Biologics Cohort (ABC) Study
Acronym: 3TR-ABC
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Bispebjerg Hospital (Other); University Hospitals, Leicester (Other); Karolinska Institutet (Other); University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof. dr. A.H. Maitland-van der Zee, Prof. Dr. Anke-Hilse Maitland- van der Zee, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 831434; ESR-21-21298 (Other Grant/Funding Number: Dutch Scientific Organization (NWO), Medical Photonics (MEDPHOT), AstraZeneca/MedImmune)
Record Dates: First submitted 2023-08-14; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Severe Asthma
Keywords: Remission; Monoclonal antibodies; Biologics
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood: 75 mL
  * Urine: 2x 80 mL (start and end of visit + urinary pellet)
  * Nasal brush: 2 nasal brushes
  * Saliva: 3 mL
  * Sputum: 3x2 mL
  * Stool: 2x 30 mL
  * BAL: 2x50 mL
  * Brush biopsies: 4
  * Mucosal biopsies: 6x50 mg, in total 300 mg
  * Skin biopsies: 2 punch skin biopsies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Severe asthma anti-IL5/IL-5R starters (including Benralizumab cohort): Patients with High dose ICS (corresponding to minimum 1600 micrograms Budesonide per day) + either LABA, LTRA, or LAMA OR Fixed Prednisolone treatment (OCS) minimum 50% of the time. Minimum 2 exacerbations in the last year or fixed Prednisolone treatment (OCS) minimum 50% of the time OR ACQ>1.5 AND Fulfils national criteria for specific biologic treatment.
- Severe asthma anti-IL4R starters: Patients with High dose ICS (corresponding to minimum 1600 micrograms Budesonide per day) + either LABA, LTRA, or LAMA OR Fixed Prednisolone treatment (OCS) minimum 50% of the time. Minimum 2 exacerbations in the last year or fixed Prednisolone treatment (OCS) minimum 50% of the time OR ACQ>1.5 AND Fulfils national criteria for specific biologic treatment.
- Severe asthma anti-TLSP starters: Patients with High dose ICS (corresponding to minimum 1600 micrograms Budesonide per day) + either LABA, LTRA, or LAMA OR Fixed Prednisolone treatment (OCS) minimum 50% of the time. Minimum 2 exacerbations in the last year or fixed Prednisolone treatment (OCS) minimum 50% of the time OR ACQ>1.5 AND Fulfils national criteria for specific biologic treatment.
- Severe asthma anti-IgE starters: Patients with High dose ICS (corresponding to minimum 1600 micrograms Budesonide per day) + either LABA, LTRA, or LAMA OR Fixed Prednisolone treatment (OCS) minimum 50% of the time. Minimum 2 exacerbations in the last year or fixed Prednisolone treatment (OCS) minimum 50% of the time OR ACQ>1.5 AND Fulfils national criteria for specific biologic treatment.
- Mild/moderate controlled asthma: Low/Medium dose of ICS/LABA +/- LTRA. ACQ < 1.5. No exacerbations in the last year or need of Prednisolone treatment (OCS). Markers of T2 inflammation (B-eos ≥ 0.15 actual or ≥ 0.30 the last year or Sputum eos ≥ 3%, FeNO ≥ 25 ppb, allergens positivity). Not direct candidate for treatments with monoclonal antibodies.
- Healthy controls: No history of respiratory diseases. No history of asthma or respiratory symptoms, normal lung function, no history of allergies. No lower or upper respiratory infections in the past 4 weeks.

SUMMARY:
The 3TR-ABC study is a multicentre observational prospective cohort study platform that follows patients with severe asthma from the start of biological therapy and three years onwards. In the 3TR-ABC platform, individual studies are conducted on specific biologics, using aligned study designs. The aim of the study is to assess response to treatment and examine clinical characteristics, biomarkers, and immunological mechanisms related to response, including remission and non-response, that might be new targets or explanations for insufficient treatment. Patients will be extensively characterized at baseline and then followed throughout the years with formal clinical and biological assessment at 4, 16, 52 weeks, and 2, 3 years. Based on the response to treatment, patients will be stratified into remission, clinical responders, and non-responders, and pre-treatment biomarker profiles obtained at the baseline visit will be compared, as well as the immunological response to treatment. Healthy individuals and patients with mild/moderate controlled asthma are included as reference groups and will undergo the same baseline visit as patients with severe asthma. Several bio-samples, to perform multi-omic analysis, will be taken to examine biological pathways associated with response and non-response to biologics.

DETAILED DESCRIPTION:
The 3TR Consortium is the overall generator behind the 3TR-ABC study. The 3TR Consortium consists of 15 European countries and a total of 69 partners who collaborate on seven different autoimmune, inflammatory, and allergic diseases: chronic obstructive pulmonary disease, asthma, Crohn's disease, ulcerative colitis, multiple sclerosis, systemic lupus erythematosus, rheumatoid arthritis. The ambition of the consortium is to accelerate precision medicine by fundamentally increasing the knowledge of molecular pathways and mechanisms related to response and non-response to therapy. To date, the 3TR Consortium is the largest immunology project funded by the Innovative Medicine Initiative (IMI). The 3TR-ABC platform study is anchored in the so-called work package 8 (WP8) within the 3TR Consortium and will contribute with knowledge about the effect of biological therapies in severe asthma: With the advent of highly targeted biological therapies for severe asthma, several important questions arise; what determines a good clinical response versus non-response? Can we induce remission of severe asthma, and improve long-term outcomes?

The 3TR-ABC study platform is a clinical trial platform and network, in which intervention-specific studies on different biologics are conducted. Via the 3TR-ABC study platform, conducting advanced translational studies in a real-life cohort of asthma patients is made possible, in collaboration with key opinion leaders and scientific experts in the field from across Europe.

The 3TR-ABC study design includes a core study visit structure, which can be expanded or amended per study to suit individual focus points.

Overall, the study design includes enrollment of bio-naïve patients with severe asthma, who have been assessed with systematic assessment, and who meet the criteria for commencing a biologic, according to national criteria in each country. Patients are then followed from the time of starting a biological treatment for three years, during which time they are followed at set time points as well as at the time of exacerbations, with sampling consisting of a core package and expanded packages, depending on the site.

By using a range of state-of-the-art and novel methods for assessing immune activation, and applying advanced bioinformatics analysis methods, The investigators expect to be able to identify immune activation patterns and response profiles that will further our understanding of disease drivers in the treatment of refractory severe asthma. Furthermore, healthy participants and patients with mild/moderate controlled asthma will be acting as controls for baseline markers thus constituting a healthy as well as mild/moderate controlled asthma reference population.

Benralizumab Cohort Study:

The AIR-BIO-OCT study Allocation to biologicals occurs by means of asthma phenotyping including clinical parameters including OCS use and blood or sputum / bronchoalveolar lavage (BAL) eosinophils (reflecting Th2 high - Th2 low inflammation). It is unclear if and how biologics impact on airway remodeling and how they act within the airway wall and which airway cells are targeted in vivo, directly or indirectly by a reduction in eosinophils. Important pathophysiological features of asthma that relate to disease severity and prognosis are airway inflammation and remodeling, including an increase in airway smooth muscle (ASM) and extracellular matrix (ECM) alterations. Therefore, with the AIR-BIO-OCT substudy as part of the 3TR-ABC Study, next to performing a complete unbiased multi-omics approach the investigators also have some already identified multi-omics phenotypes within severe asthma that the investigators would like to investigate in a cohort of benralizumab users. As such extensive phenotyping before and after treatment, by combining exhaled breath VOCs (GC-MS and eNose) technology with minimal invasive omics (molecular) and innovative imaging technology by OCT, including polarization-sensitive OCT PS-OCT (impact of benralizumab on remodeling).

Primary Objective Determine baseline biomarkers of remission after 1 year of biological therapy, defined as ACQ-5 <1.5, post-bronchodilator FEV1 percent predicted ≥80% OR >10% improvement as well as no exacerbations, or use of maintenance steroids for the past 12 months ("remission on treatment").

Secondary Objectives Determine baseline biomarkers of remission after 3 years of biological therapy. Additionally, i) Change in biomarker profiles in remission versus non-remission groups, ii) baseline and change in biomarker profile for a) each response outcome individually, b) Global evaluation treatment efficacy (GETE), patient and physician rated response, and c) 3TR agreed on a composite assessment of response, iii) determine the change in all response variables against baseline biomarker data and change in biomarkers as continuous variables.

Exploratory Objectives: Novel analytical science approaches including but not limited to network and cluster analyses and partial least-squared discriminate analysis (PLSDA), topographical discriminant analysis of omic data derived from the biosamples collected at planned visits as well as daily FENO to determine possible novel biomarker signatures (including FENO) and relate to asthma remission, clinical response, interactomes of the multi-omic and clinical data, host-microbiome interactions.

AIR-BIO-OCT substudy objectives

Primary Objective:

* To identify and measure an eNose/ volatile organic compound (VOC)- multi-omics extensive severe asthma phenotyping strategy before treatment with biologicals to reveal add-on response characteristics to better predict treatment response.
* To identify and measure minimal invasive predicting "signature" of biological treatment response in severe eosinophilic asthma by extensive asthma pheno-endotyping using innovative minimal invasive exhaled breath technologies including eNose/VOCs and omics.

Secondary Objective(s)

* To measure airway remodeling (extracellular matrix and airway smooth muscle) after treatment with Benralizumab
* Establish the reduction of extracellular matrix (ECM) and airway smooth muscle (ASM) by the standard - polarization-sensitive (PS) - OCT and endobronchial biopsy analyses after 6 months - 1 year of Benralizumab treatment.

Study Design

The 3TR-ABC study is a multicentre observational prospective cohort study that follows patients with severe asthma from the time of commencement of biological therapy and three years onwards.

Healthy individuals and patients with mild/moderate controlled asthma are included as reference groups and will undergo the same baseline visit as patients with severe asthma.

Informed Consent must be obtained from all participants who accept enrollment in the study in order to allow the collection of data and biological materials for the database and biobank, respectively.

The study follows each patient with severe asthma at six visits over a period of three years. The first visit is the so-called baseline visit and is performed before the beginning of a biological treatment. This visit consists of a standard examination package, a site-specific extended package (i.e., tests in this package will only be done at specific sites), and an optional extended package (i.e., the participant decides). The remaining five visits are so-called follow-up visits and are made respectively 4 weeks, 16 weeks, 52 weeks, 2 years, and 3 years after the baseline visit. These visits consist of a follow-up sampling package and a site-specific extended package. An optional extended package is furthermore possible for the 4 weeks, 52 weeks, 2 years, and 3 years visits. Between scheduled visits, patients with severe asthma are asked to come for an extra visit if they experience a sudden exacerbation. Participants in the control groups will only be invited for the baseline visit.

The AIR-BIO-OCT study is a sub-study within the 3TR-ABC Study performed in the Netherlands that will select severe eosinophilic asthma patients that start treatment with Benralizumab and will phenotype those patients (combining exhaled breath analysis and OCT technology) before and after 16 weeks and additional 52 weeks from the start of the biological. In the Netherlands, the AIR-Bio-OCT substudy consists of two parts: the first, aligned with the 3TR - ABC study, where samples of the abovementioned packages will be collected (n=34) and merged with the Benralizumab subjects recruited within the 3TR consortium (total 60-90 patients). The second part, additional bronchoscopy with standard and PS-OCT before and after 6 months-1 year will be performed (n=15).

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe asthma that requires High dose ICS (corresponding to minimum 1600 micrograms Budesonide per day) + either LABA, LTRA, or LAMA OR Fixed Prednisolone treatment (OCS) minimum 50% of the time. Minimum 2 exacerbations in the last year or fixed Prednisolone treatment (OCS) minimum 50% of the time OR ACQ>1.5 AND Fulfils national criteria for specific biologic treatment.
* Patients with mild/moderate asthma that requires Low/Medium dose of ICS/LABA +/- LTRA. ACQ < 1.5. No exacerbations in the last year or need of Prednisolone treatment (OCS). Markers of T2 inflammation (B-eos ≥ 0.15 actual or ≥ 0.30 the last year or Sputum eos ≥ 3%, FeNO ≥ 25, allergens positivity). Not direct candidate for treatments with monoclonal antibodies.
* Healthy volunteers that reports no respiratory diseases, No history of asthma or respiratory symptoms, normal lung function. No history of allergies. No lower or upper respiratory infections in the past 4 weeks.

Exclusion Criteria:

* Patients with severe asthma:

  1. Known hypersensitivity to the active substance or any of the excipients
  2. Participation in an interventional clinical trial within 3 months of visit 1 or receipt of any investigational medicinal product within 3 months or 5 half-lives. Participation in other observational studies is acceptable if in the view of the investigator it will not impact on the study outcomes.
  3. Other clinically significant medical disease or uncontrolled concomitant disease that is likely, in the opinion of the investigator, to require a change in therapy or impact the ability to participate in the study.
* Patients with mild/moderate asthma:

  1. Unable to understand written information due to language barriers.
  2. Unable to give informed consent, i.e., patients who are incapable.
  3. Show sign of symptoms of uncontrolled asthma (ACQ score higher than 1.5, OCS use, history of exacerbations within the past year).
* Healthy volunteers:

  1. Unable to understand written information due to language barriers.
  2. Unable to give informed consent, i.e., patients who are incapable.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will constitute a real-life population of patients with severe asthma, who are eligible to receive biological treatment according to relevant national criteria. The study will include all age groups.
  Furthermore, the study will include two control groups, a group of mild/moderate asthmatics and a group of healthy volunteers. All controls will be age-, sex-, and smoking-history-matched with the group of patients with severe asthma. The rationale behind the control groups is to compare those patients who show the best response to Anti-IgE, Anti-IL5(R), Anti-IL4/IL13, anti-TSLP treatments with those who are not candidate for a biologic therapy, both mild/moderate asthmatics and healthy individuals. In this way, the study aims to explore whether there are biomarkers indicative of a better response to monoclonal antibodies.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2033-08 (Estimated)

PRIMARY OUTCOMES:
Change in Asthma Control Questionnaire 5 (ACQ-5) score | 1 year, 2 and 3 years
  This is a validated score that includes 5 questions scored from 0 to 6 with the total score being the average of the questions. The ACQ score ranges between 0 (well controlled) and 6 (extremely poorly controlled). A score of 1.5 or more indicates that a patient has inadequate asthma control.
Change in post- broncodilator Forced Expiratory Volume after 1 second (FEV1) | 1 year, 2 and 3 years
  This is a validated parameter, part of regular clinical care, to assess airway obstruction using a spirometry. A dose of bronchodilator medication is administered by means of inhaler or nebulizer (such as 400mcg of salbutamol). and the spirometry is repeated after 15 minutes. An increase of the FEV1 >10% compared to the baseline or a FEV1 ≥80% indicates good asthma control
Absense of exacerbations | 1 year, 2 and 3 years
  Asthma exacerbations are acute or subacute episodes of progressively worsening shortness of breath, cough, wheezing, and chest tightness-or some combination of these symptoms.
No usage of oral corticosteroids in the previous 12 months | 1 year, 2 and 3 years
  Oral corticosteroids (OCS) are a common treatment for acute asthma flare-ups to reduce inflammation and swelling in the airways. Severe asthma patients can be oral corticosteroids dependent and the reduction of the usage of oral corticosteroids will indicate a good asthma control.

SECONDARY OUTCOMES:
Change in volatile organic compounds (VOC) | 1, 2, 3 years
  VOCs are exhaled during normal breathing to reflect potential pathophysiological changes of the airways. The concentration of the compounds with breath will be measure using Gas chromatography-mass spectrometry (GC-MS).
Measure airway remodeling | 6 months to 1 year of benralizumab treatment
  The reduction of extra cellular matrix (ECM) and/of airway smooth muscle (ASM) by standard -using a new technique, the polarization sensitive (PS) - OCT and endobronchial biopsy analyses

OTHER OUTCOMES:
Variability of Fraction Exhaled Nitric Oxide (FeNO) | 3 years
  This validated test is performed using a portable device that measures the level of nitric oxide in parts per billion (PPB) in the air slowly exhaled out of lungs.

CONTACTS AND LOCATIONS:
Overall Officials: Anke-Hilse Maitland-van der Zee, Prof.Dr., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Peter Bonta, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Celeste Porsbjerg, Prof.Dr., Principal Investigator — Bispebjerg Hospital; Christopher E. Brightling, Prof. Dr., Principal Investigator — University of Leicester; Sven-Erik Dahlén, Prof. Dr., Principal Investigator — Karolinska Intitutet
Locations (2):
- Bispebjerg Hospital, Copenhagen, Denmark
- Amsterdam University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided